CLINICAL TRIAL: NCT03954470
Title: Factors Influencing Risk of Progression of Chronic Kidney Disease in Patients With Severe Renal Failure
Brief Title: Factors Influencing Risk of Progression of Chronic Kidney Disease
Acronym: FAIR-PROGRESS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2017/87
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Chronic Kidney Disease stage4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify typical patterns of renal function evolution in patients with stage 4 chronic kidney disease, regularly followed in nephrology consultation and included in a French cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the inclusion criteria of the ND-CRIS cohort (long-term follow-up in one of the centers participating in the research, with a GFR <60mL/min /1.73m2)
* Patients included in the ND-CRIS cohort on the date when the estimate of their GFR is strictly less than 30mL/min/1.73m2 and greater than or equal to 15mL/min/1.73m2 (MDRD equation).

Patients should have at least two measurements of GFR <30mL/min/1.73m2 to be included, at least one of them greater than or equal to 15mL/min/1.73m2. The date of the first GFR <30mL/min/ 1.73m2 will be considered as the date of origin.

Exclusion Criteria:

* Patients with GFR ≥30mL / min / 1.73m2 or <15mL / min / 1.73m2
* Patients who do not meet the inclusion criteria of ND-CRIS cohort (dialysis patients, transplant patients, unfollowed patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with chronic renal failure, before replacement therapy, followed in 9 nephrology departments of Bourgogne Franche-Comté.
Sampling Method: Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2012-04-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evolution of estimated Glomerular Filtration Rate (GFR) according to MDRD equation (modification of diet in renal disease) at each visit | up to 3 years
Time between inclusion and occurrence of the "progression" event | up to 3 years
  progression: initiation of an extra-renal purification technique or reduction of GFR of at least 5 mL / min / 1.73m2 compared to inclusion in FAIR-PROGRESS

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France